## Post Excision/Mohs Fractional CO2 Resurfacing: A Quantitative and Qualitative Scar Analysis Study PI: Hooman Khorasani NCT02130297

Document Date: 3/9/18

Post Excision/Mohs Fractional CO2 Resurfacing: A Quantitative and Qualitative Scar Analysis Study

11 Quantitative and Quanta

PI: Hooman Khorasani, MD

**Date**: 3/9/18

Statistical analyses

The scars were assessed 6 months after surgery. Each subject was asked if one scar half appeared

cosmetically better than the other or if both halves looked cosmetically equivalent. A physician, blinded

to treatment, then assessed each half of the scar according to the validated modified Manchester scar

scale (MMSS).16

3mm punch biopsies were then extracted from each scar half and subjected to quantitative scar

analysis. Biopsies were fixed in formalin then dehydrated, paraffin-embedded and breadloafed into

sections for picrosirius red staining. For analysis of collagen architecture, confocal photographs were

captured by a Leica<sup>©</sup> TCSSPMP confocal microscope (Leica Microsystems<sup>©</sup>, Wetzlar, Germany) at 1000

fold magnification.<sup>17</sup> Sections were scanned in 1 micron increments for the entire section thickness of 7

microns. Data of frame-mode images were recorded and stored as 512 pixel images. Fractal dimension

(F<sub>D</sub>) and lacunarity (L) analyses were performed on the confocal images using a previously described

methodology.<sup>18</sup>

This method for quantitative scar analysis was chosen because confocal microscopy leverages the

fluorescence properties of collagen and provides high resolution images of dermal structure. Scar tissue

exhibits denser (higher F<sub>D</sub>) and more homogenous (lower L) architecture compared with the looser,

basket-weave pattern of normal skin. It, therefore, follows that cosmetically superior scar tissue should

closely resemble normal skin, with a lower F<sub>D</sub> and higher L. Pairwise t-test comparison was performed using Stata® 12 software (StataCorp LLC, College Station, Texas).